CLINICAL TRIAL: NCT00671333
Title: A Randomized Prospective Study Comparing Ligament Reconstruction and Tendon Interposition (LRTI) With a Joint Spacer (Ascension PyroDisk) for Trapeziometacarpal Osteoarthritis.
Brief Title: PRCT: Ligament Reconstruction & Tendon Interposition With a Joint Spacer for Trapeziometacarpal OA
Acronym: TMC/PyroDisk
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study fatigue
Sponsor: Fraser Orthopaedic Research Society (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-060
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Joint Disease
Keywords: Randomized; Prospective; Procedure / Surgery
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): (LRTI) Ligament reconstruction and tendon interposition
  Interventions: Procedure: LRTI
- 2 (Active Comparator): Ascension PyroDisk
  Interventions: Procedure: Ascension PyroDisk

INTERVENTIONS:
Procedure: LRTI — Dorsal radial incision, capsulotomy between EPB and APL protecting the radial artery, trapeziectomy using a cruciate osteotomy and rongeurs, creation of a metacarpal base bone tunnel using a high speed burr, harvesting of entire FCR tendon through two transverse volar incisions, ligament reconstruction and tendon interposition using "Fibre Wire" suture. Closure of capsule with Vicryl. Closure of skin with running Prolene suture.
  Arms: 1
Procedure: Ascension PyroDisk — Dorsal radial incision, capsulotomy between EPB and APL protecting the radial artery, distal 2 mm of trapezium and dorsal cortex of both trapezium and metacarpal removed using osteotomes/rongeurs. A hole is drilled through the trapezium from dorsal to resected distal surface, and a second hole is drilled through the first metacarpal from the resected base to the dorsal surface. A slip of FCR is harvested. The tendon is woven through the trapezium, the central hole in the device, and the metacarpal tunnel then sutured back onto itself. Closure of capsule with Vicryl. Closure of skin with running Prolene suture.
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effectiveness of two types of operative treatment in terms of resolving symptoms, improving function and also with respect to x-ray outcomes.

The hypothesis is that insertion of a spacer will provide similar symptomatic relief, but improved long term gains in key and tripod pinch strength when compared to LRTI.

DETAILED DESCRIPTION:
Trapeziometacarpal (TMC) arthritis is a common condition, which occurs when the cartilage (tissue) covering the bones at the joint at the base of the thumb wear away. This condition occurs in 10% of women and 1% of men.

There is controversy regarding the best treatment of this condition and many surgical techniques are in common use.

One of these involves removing the wrist bone (trapezium) at the base of the thumb and, using a tendon from the forearm, reconstructing an important ligament, which contributes to the stability of the thumb. This is known as a Ligament Reconstruction and Tendon Interposition (LRTI).

A newer type of operation involves the insertion of a Ascension PyroDisk which is made from a thick pyrocarbon layer encasing a graphite core with a small amount of tungsten. These materials have been shown to be safe when implanted in the body. The PyroDisk is a disk shaped design which has a curved surface designed to fit between the bony surfaces of the trapezium and the metacarpal, reducing pain and allowing for full movement of the joint. It contains a hole in the center through which a strip of tendon can be passed and helps hold the disk in place.

This research study is designed to determine the effectiveness of the Ascension PyroDisk spacer when compared to the LRTI procedure described above. The effectiveness of both of these procedures will be determined by comparing range of motion, grip and pinch strength, x-rays, function and return to work. It is important to compare both procedures, as it is not known which procedure is the most effective.

ELIGIBILITY:
Inclusion Criteria:

* isolated trapeziometacarpal osteoarthritis
* duration of symptoms of at least six months
* failure to respond to non-operative management
* age 50 or older
* less than 30 degrees of ipsilateral MCP hyperextension
* British Columbian resident living in the Lower Mainland and available for protocol follow-up

Exclusion Criteria:

* previous surgery for TMC arthritis
* other significant ipsilateral wrist or hand pathology
* a history of inflammatory arthropathy
* a requirement for concommitant surgery for another condition
* any previous hand or wrist fracture

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2008-04; Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
Patient Rated Wrist Evaluation (PRWE) at baseline, 6 weeks, 3, 6 and 12 months post-operatively. | Subjects are followed for 12 months post-op.

SECONDARY OUTCOMES:
Wrist range of motion, grip strength, radiographs, and pain Visual Analog Scale. | Baseline, 6 weeks, 3,6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand H Perey, MD, Principal Investigator — Royal Columbian Hospital, Eagle Ridge Hospital
Locations (2):
- Canada (2):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Eagle Ridge Hospital, Port Moody, British Columbia

REFERENCES:
- [Background] Armstrong AL, Hunter JB, Davis TR. The prevalence of degenerative arthritis of the base of the thumb in post-menopausal women. J Hand Surg Br. 1994 Jun;19(3):340-1. doi: 10.1016/0266-7681(94)90085-x. PMID 8077824
- [Background] Eaton RG, Littler JW. Ligament reconstruction for the painful thumb carpometacarpal joint. J Bone Joint Surg Am. 1973 Dec;55(8):1655-66. No abstract available. PMID 4804988
- [Background] Wilson JN, Bossley CJ. Osteotomy in the treatment of osteoarthritis of the first carpometacarpal joint. J Bone Joint Surg Br. 1983 Mar;65(2):179-81. doi: 10.1302/0301-620X.65B2.6826626.
- [Background] Carroll RE, Hill NA. Arthrodesis of the carpo-metacarpal joint of the thumb. J Bone Joint Surg Br. 1973 May;55(2):292-4. No abstract available. PMID 4707297
- [Background] Burton RI, Pellegrini VD Jr. Surgical management of basal joint arthritis of the thumb. Part II. Ligament reconstruction with tendon interposition arthroplasty. J Hand Surg Am. 1986 May;11(3):324-32. doi: 10.1016/s0363-5023(86)80137-x. PMID 3711604
- [Background] GERVIS WH. Excision of the trapezium for osteoarthritis of the trapezio-metacarpal joint. J Bone Joint Surg Br. 1949 Nov;31B(4):537-9, illust. No abstract available. PMID 15397137
- [Background] Swanson AB. Disabling arthritis at the base of the thumb: treatment by resection of the trapezium and flexible (silicone) implant arthroplasty. J Bone Joint Surg Am. 1972 Apr;54(3):456-71. No abstract available. PMID 5055148
- [Background] Cooney WP, Linscheid RL, Askew LJ. Total arthroplasty of the thumb trapeziometacarpal joint. Clin Orthop Relat Res. 1987 Jul;(220):35-45. PMID 3595008
- [Background] Tomaino MM, Pellegrini VD Jr, Burton RI. Arthroplasty of the basal joint of the thumb. Long-term follow-up after ligament reconstruction with tendon interposition. J Bone Joint Surg Am. 1995 Mar;77(3):346-55. doi: 10.2106/00004623-199503000-00003. PMID 7890782
- [Background] Low AK, Edmunds IA. Isolated scaphotrapeziotrapezoid osteoarthritis: preliminary results of treatment using a pyrocarbon implant. Hand Surg. 2007;12(2):73-7. doi: 10.1142/S0218810407003523. PMID 18098356
- [Background] Nunez VA, Citron ND. Short-term results of the Ascension pyrolytic carbon metacarpophalangeal joint replacement arthroplasty for osteoarthritis. Chir Main. 2005 Jun-Aug;24(3-4):161-4. doi: 10.1016/j.main.2005.04.009. PMID 16121621
- [Background] Heers G, Grifka J, Borisch N. [First results after implantation of a pyrocarbon-endoprosthesis in patients with degenerative arthritis]. Z Orthop Ihre Grenzgeb. 2006 Nov-Dec;144(6):609-13. doi: 10.1055/s-2006-955189. German. PMID 17187336
- [Background] Beckenbaugh RD. [Arthroplasty of the metacarpophalangeal joint using pyrocarbonate implants]. Orthopade. 2003 Sep;32(9):794-7. doi: 10.1007/s00132-003-0519-x. German. PMID 14508645